CLINICAL TRIAL: NCT00208715
Title: A DOUBLE-BLIND PILOT STUDY TO EVALUATE THE SAFETY AND EFFICACY OF PROVIGIL® (MODAFINIL) AT FIXED/FLEXIBLE DOSES, IN CONJUNCTION WITH IDENTIFIED SSRIs FOR THE TREATMENT OF EXCESSIVE SLEEPINESS IN PATIENTS WITH MILD TO MODERATE DEPRESSION WITH ATTENDANT SYMPTOMS OF SLEEPINESS AND FATIGUE
Brief Title: Provigil in Conjunction With SSRIs for the Treatment of Mild or Moderate Depression With Attendant Symptoms of Sleepiness and Fatigue.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1021-2002
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Major Depression; Mental Health
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression | interventions — Modafinil

INTERVENTIONS:
Drug: Provigil

SUMMARY:
The main purpose of this study is to determine if Provigil® (modafinil) at a dose of 200 mg once daily is safe and effective for treating symptoms of sleepiness and fatigue associated with Major Depressive Disorder when added to a SSRI.

DETAILED DESCRIPTION:
Approximately 100 male and female outpatients, who are between the ages of 18 and 65, will be enrolled at four sites in the United States. This study consists of two parts. The first part consists of 6 weeks of open label treatment with a selected SSRI & double blind treatment with Provigil or placebo (inactive medication).

After the six week double blind treatment phase all patients will enter a four week open label treatment phase with Provigil. The dose of Provigil is not to exceed 400 mg and cannot be less than 100 mg per day. They will continue taking the prescribed SSRI.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* MADRS score ≥ 15 at both screen & baseline.
* Significant fatigue as evidenced by FSS ≥4 at both screen & baseline.
* Excessive sleepiness as evidenced by ESS ≥ 10 at both screen & baseline.

Exclusion Criteria:

* Treatment refractory depression
* Serious or unstable medical condition.
* Pregnancy
* Primary diagnosis of another Axis I or II disorder
* Alcohol or substance abuse or dependence within the past 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-02; Study Completion 2004-10

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS)

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAM-D 31 item)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Ninan, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania